CLINICAL TRIAL: NCT04679077
Title: Preoperative Microcirculation and Postoperative Outcome After Major Vascular Surgery: a Prospective Cohort Study
Brief Title: Preoperative Microcirculation and Postoperative Outcome After Major Vascular Surgery
Acronym: MAPOVAS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was never submitted to the ethics committee
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MAPOVAS
Record Dates: First submitted 2020-12-09; First posted 2020-12-22 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Surgery--Complications

STUDY DESIGN:
Intervention Model Description: Patients will be split into two groups after data collection. They will receive the same treatment during the clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cytocam-IDF Imaging (Other): All patients will undergo the same interventional test.
  Interventions: Other: Cytocam-IDF imaging device

INTERVENTIONS:
Other: Cytocam-IDF imaging device — Observation of the microcirculation

SUMMARY:
The aim of the study is to determine whether there is a correlation between the microcirculation measured preoperatively in patients undergoing major vascular surgery and the postoperative mortality during hospitalization period. The microcirculation will be measured sublingually with the Cytocam-IDF imaging technique.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years

  * Males and females
  * ASA III classification
  * Written informed consent obtained by the patient
  * Elective hospital admission for major vascular surgery, both open and endovascular

Exclusion Criteria:

* Emergency surgery

  * Minor vascular procedures (e.g. varicose vein stripping; thromboembolectomy; vascular access formation)
  * Pregnancy
  * Refusal or inability to provide written informed consent (language barrier, mental retardation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative high-sensitive troponin T (hsTnT) | 30 days
  Indicator of acute coronary syndrome

SECONDARY OUTCOMES:
Cause of death | 30 days
  Causes of death
Non-cardiovascular adverse events and serious adverse events | 30 days
  Incidence of non-cardiovascular complications
Cardiovascular adverse events and serious adverse events | 30 days
  Incidence of cardiovascular complications
Correlation between preoperative microcirculation and postoperative outcome during the hospitalization period. | 30
  In addition, demographic parameters (age, weight, height) and comorbidities will be taken into account.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
Presentations of both the study protocol and the study results will be held at conferences.
  After completion of the study and analysis of the data results will be made publicly without re striction, independent of the outcome. They will be submitted for publication to an international peer-reviewed journal.